CLINICAL TRIAL: NCT02658851
Title: Application of Cold Plasma Energy for Reduction of Lymphoceles Following Pelvic Lymph Node Dissection During Robot-Assisted Radical Prostatectomy
Brief Title: Cold Plasma for the Reduction of Lymphoceles Following PLND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 808076
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Lymphoceles Following Pelvic Lymph Node Dissection
Keywords: lymphocele; pelvic lymph node dissection; robotic assisted radical prostatectomy; PLND; RARP; prostatectomy; Patel
MeSH Terms: conditions — Lymphocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- J-Plasma (Experimental): Enrolled participants will have their PLND performed using J-Plasma® for dissection and sealing of lymphatic channels.
  Interventions: Device: J-Plasma

INTERVENTIONS:
Device: J-Plasma — Bovie Medical Corporation's J-Plasma® helium based plasma technology is a hemostatic tool for the cutting, coagulation, and ablation of soft tissue.
  Other Names: Cold plasma

SUMMARY:
This study protocol will evaluate the efficacy of Bovie Medical's J-Plasma® helium based plasma technology in the reduction of lymphoceles following pelvic lymph node dissection (PLND) during robotic assisted radical prostatectomy (RARP). The J-Plasma® handpiece will be used during the PLND by dissecting the lymph nodes and sealing the lymphatic channels to prevent lymph leakage.

DETAILED DESCRIPTION:
Participants evaluated and scheduled for a PLND during Robotic Assisted Radical Prostatectomy who have met the study inclusion criteria and who have also given informed consent will be enrolled. Enrolled participants will have their PLND performed using J-Plasma® for dissection and sealing of lymphatic channels. An abdominal-pelvic ultrasound will be completed at a follow-up period ranging from 4-12 weeks post operatively to determine if a lymphocele is present. The occurrence rate of lymphoceles in this trial group will be compared to retrospective data from the principal investigator's practice and other published data to determine if the occurrence rate has been reduced.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of Prostate Cancer (ICD-10:C61)
2. Prostate Specific Antigen (PSA) level =/> 10ng/mL
3. Gleason score =/> 7
4. Planned Elective Robotic Assisted Radical Prostatectomy with planned pelvic lymph node dissection.
5. Willing and able to return to clinic for standard of care abdominal ultrasound within 12 weeks post operatively.
6. Able to provide informed consent

Exclusion Criteria:

Must answer no to all:

1. Patient is unwilling or unable to sign or understand informed consent
2. Patient resides outside of the United States
3. Performance of Lymph node dissection was aborted.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vipul R Patel, MD, Principal Investigator — Florida Hospital Global Robotics Institute
Locations (1):
- Florida Hospital Global Robotics Institute, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | J-Plasma
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | J-Plasma
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.28 (7.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 83
  More than one race | 0
  Unknown or Not Reported | 3
Pre-Op Prostate-Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 7.97 (5.23)
Pre-Operative Biopsy Gleason [Mean (Standard Deviation); unit: units on a scale (Scale 2 - 10)] — Gleason scores range from 2 to 10, and most prostate cancer will score 6 or higher. A higher score (8 to 10) means the type of cancer has a higher risk of growing and spreading.
  units on a scale (Scale 2 - 10) | 7.45 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Lymphocele Formation
Description: The primary outcome to be measured will be the incidence of lymphocele formation as diagnosed upon post- operative abdominal ultrasound.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | J-Plasma
Number analyzed (Participants) | 100
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at the day of surgery and collected to the 8 week follow-up visit (8 weeks, +/- 4 weeks)
Arm/Group | J-Plasma
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT02658851/Prot_SAP_000.pdf